CLINICAL TRIAL: NCT05101252
Title: Comparison of a Daily Disposable Multifocal Contact Lens to a Marketed Product
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johnson & Johnson Vision Care, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CR-6468
Record Dates: First submitted 2021-10-08; First posted 2021-11-01 (Actual); Results first posted 2023-01-10 (Actual); Last update posted 2023-01-10 (Actual); Status verified 2022-12

CONDITIONS: Visual Acuity

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- TEST Lens (Active Comparator): Eligible subjects who are habitual soft contact lens wearers will be randomized to the TEST Lens sequence for the duration of the study.
  Interventions: Device: senofilcon A C3
- CONTROL Lens (Experimental): Eligible subjects who are habitual soft contact lens wearers will be randomized to the CONTROL Lens sequence for the duration of the study.
  Interventions: Device: Dailies Total 1 Multifocal Contact Lenses

INTERVENTIONS:
Device: senofilcon A C3 — TEST Lens
  Arms: TEST Lens
Device: Dailies Total 1 Multifocal Contact Lenses — CONTROL Lens
  Arms: CONTROL Lens

SUMMARY:
This is a single-masked, two-arm, parallel-group, randomized-controlled, dispensing clinical trial to evaluate the visual performance.

ELIGIBILITY:
Inclusion Criteria:

* Potential subjects must satisfy all the following criteria to be enrolled in the study:

  1. Read, understand, and sign the STATEMENT OF INFORMED CONSENT and receive a fully executed copy of the form.
  2. Appear able and willing to adhere to the instructions set forth in this clinical protocol.
  3. Be at least 40 years of age and not greater than 70 years of age at the time of consent.
  4. Own a wearable pair of spectacles if required for their distance vision.
  5. Be an adapted soft contact lens wearer in both eyes (i.e. worn lenses a minimum of 2 days per week for at least 6 hours per wear day, for 1 month or more duration).
  6. Either already be wearing a presbyopic contact lens correction (e.g., reading spectacles over contact lenses, multifocal or monovision contact lenses, etc.) or if not respond positively to at least one symptom on the "Presbyopic Symptoms Questionnaire".
  7. The subject's distance spherical equivalent refraction must be in the range of -1.25 D to -3.75 D or +1.25 D to +3.75 D in each eye.
  8. The subject's refractive cylinder must be ≤0.75 D in each eye.
  9. The subject's ADD power must be in the range of +0.75 D to +2.50 D.
  10. The subject must have distance best corrected visual acuity of 20/20-3 or better in each eye.

      Exclusion Criteria:
* Potential subjects who meet any of the following criteria will be excluded from participating in the study:

  1. Be currently pregnant or lactating.
  2. Have any active or ongoing ocular or systemic allergies that may interfere with contact lens wear.
  3. Have any active or ongoing systemic disease, autoimmune disease, or use of medication, which may interfere with contact lens wear. This may include, but not be limited to, diabetes, hyperthyroidism, Sjögren's syndrome, xerophthalmia, acne rosacea, Stevens-Johnson syndrome, and immunosuppressive diseases or any infectious diseases (e.g. hepatitis, tuberculosis).
  4. Have any previous, or planned, ocular or intraocular surgery (e.g. radial keratotomy, PRK, LASIK, lid procedures, cataract surgery, retinal surgery, etc.).
  5. Have a history of amblyopia, strabismus or binocular vision abnormality.
  6. Use of any of the following medications within 1 week prior to enrollment: oral retinoid, oral tetracyclines, anticholinergics, oral phenothiazines, oral/inhaled corticosteroids. See Table 9.1 for further examples.
  7. Use of any ocular medication, with the exception of rewetting drops.
  8. Have a history of herpetic keratitis.
  9. Have a history of irregular cornea.
  10. Have a history of pathological dry eye.
  11. Have Participated in any contact lens or lens care product clinical trial within 30 days prior to study enrollment.
  12. Be and employee or immediate family member of an employee of clinical site (e.g., Investigator, Coordinator, Technician).
  13. Have any known hypersensitivity or allergic reaction to non-preserved rewetting drop solutions or sodium fluorescein.
  14. Have clinically significant (Grade 3 or greater) corneal edema, corneal vascularization, corneal staining, tarsal abnormalities or bulbar injection, or any other corneal or ocular abnormalities which would contraindicate contact lens wear.
  15. Have any current ocular infection or inflammation.
  16. Have any current ocular abnormality that may interfere with contact lens wear.

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 77 (Actual)
Dates: Start 2021-10-11 (Actual); Primary Completion 2021-11-29 (Actual); Study Completion 2021-11-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Vision Care, Inc. Clinical Trial, Study Director — Johnson & Johnson Vision Care, Inc.
Locations (9):
- United States (9):
  - Stam & Associates Eye Care, Jacksonville, Florida
  - Sabal Eye Care, Longwood, Florida
  - Visual Eyes, Roswell, Georgia
  - Kannarr Eye Care, Pittsburg, Kansas
  - Birmingham Vision Care, Bloomfield Township, Michigan
  - Eye Associates of New York, New York, New York
  - ProCare Vision Centers, Granville, Ohio
  - West Bay Eye Associates, Warwick, Rhode Island
  - Tyler Eye Associates, Tyler, Texas

IPD SHARING:
Plan to Share IPD: Yes
Johnson & Johnson Medical Device Companies have an agreement with the Yale Open Data Access (YODA) to serve as the independent review panel for evaluation of requests for clinical study reports and participant level data from investigators and physicians for scientific research that will advance medical knowledge and public health. Requests for access to the study data can be submitted through the YODA Project site at http://yoda.yale.edu
URL: http://yoda.yale.edu

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 77 subjects were enrolled in this study. Of those enrolled, 74 subjects were dispensed at least one study lens, while 3 subject failed to meet all eligibility criteria. Of those dispensed, 69 subjects completed the study while 5 subjects were discontinued.
Groups:
- Test (Senofilcon A C3): Subjects that wore the Test lens during the study.
- Control (Delefilcon A): Subjects that wore the Control lens during the study.
Period: Overall Study
Arm/Group | Test (Senofilcon A C3) | Control (Delefilcon A)
Started | 37 | 37
Completed | 35 | 34
Not Completed | 2 | 3
Not completed — Unsatisfactory Test Article | 1 | 0
Not completed — Subject Withdrawn by PI due to Non Compliance to Protocol | 0 | 1
Not completed — Withdrew Consent during study | 0 | 1
Not completed — Subject dispensed incorrect lens in 1 eye | 1 | 1

BASELINE CHARACTERISTICS:
Population: All subjects dispensed a study lens with data collected at the 1-week follow-up evaluation.
Groups:
- Total: Total of all reporting groups
Arm/Group | Test (Senofilcon A C3) | Control (Delefilcon A) | Total
Number analyzed (Participants) | 36 | 34 | 70
Age, Continuous [Mean (Standard Deviation); unit: Years] | 58.0 (5.95) | 55.4 (5.48) | 56.7 (5.84)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 31 | 24 | 55
  Male | 5 | 10 | 15
Race/Ethnicity, Customized [Number; unit: Participants]
  Asian | 1 | 1 | 2
  Black or African American | 3 | 3 | 6
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  White | 32 | 29 | 61
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 36 | 34 | 70

OUTCOME MEASURES:

1. Primary Outcome: Binocular logMAR Visual Acuity
Description: Binocular visual acuity was measured on a logMAR (Logarithm of Minimal Angle of Resolution) scale under high luminance high contrast condition. At distance (4 meters), VA is assessed using ETDRS (Early Treatment Diabetic Retinopathy Study) charts; while near (40 cm) and intermediate (64 cm) assessments were made using reduced Guillon-Poling charts. Letter-by-letter results calculated the visual performance score for each chart read. LogMAR scores closer to zero, or below zero, indicate a better visual acuity. A logMAR visual performance score of 0.0 is equivalent to Snellen visual acuity of 20/20.
Time Frame: 1-Week Follow-up
Population: All randomized subjects regardless of actual treatment and subsequent withdrawal from study or deviation from protocol, with data at the 1-Week Follow-up Evaluation.
Measure: Mean (Standard Deviation); unit: LogMAR
Arm/Group | Test (Senofilcon A C3) | Control (Delefilcon A)
Number analyzed (Participants) | 36 | 34
LogMAR
  Distance (4m) | -0.076 (0.0915) | -0.081 (0.1052)
  Intermediate (64cm) | 0.006 (0.0876) | -0.013 (0.0934)
  Near (40cm) | 0.090 (0.0924) | 0.084 (0.0904)
Statistical Analysis 1: Comparison: Test (Senofilcon A C3); It was calculated using a 2-sided one sample mean t-test with a family wise type I error rate of 5% (1.25% individually) with at least 90% statistical power, that 22 subjects were required to test for superiority for distance; Test type: Superiority — Superiority was declared if the upper limit of the 98.75% confidence interval of was below 0.00 logMAR for distance; Linear Mixed Model; Kenward and Roger method was used for denominator degrees of freedom; Least-square Mean = -0.08, 98.75% CI 2-sided [-0.14 to -0.01], Standard Error of Mean 0.022
Statistical Analysis 2: Comparison: Test (Senofilcon A C3); It was calculated using a 2-sided one sample mean t-test with a family wise type I error rate of 5% (1.25% individually) with at least 90% statistical power, that 12 subjects were required to test for superiority for intermediate; Test type: Superiority — Superiority was declared if the upper limit of the 98.75% confidence interval of was below 0.17 logMAR for intermediate; Linear Mixed Model; Kenward and Roger method was used for denominator degrees of freedom; Least-square Mean = 0.00, 98.75% CI 2-sided [-0.06 to 0.07], Standard Error of Mean 0.022
Statistical Analysis 3: Comparison: Test (Senofilcon A C3); It was calculated using a 2-sided one sample mean t-test with a family wise type I error rate of 5% (1.25% individually) with at least 90% statistical power, that 60 subjects were required to test for superiority for near; Test type: Superiority — Superiority was declared if the upper limit of the 98.75% confidence interval of was below 0.17 logMAR for near; Linear Mixed Model; Kenward and Roger method was used for denominator degrees of freedom; Least-square Mean = 0.09, 98.75% CI 2-sided [0.02 to 0.16], Standard Error of Mean 0.023

2. Primary Outcome: CLUE Vision Score
Description: Subjective vision was assessed using the Contact Lens User Experience™ (CLUE) questionnaire. CLUE is a validated patientreported outcomes (PRO) questionnaire to assess patient-experience attributes of soft contact lenses (comfort, vision, handling, and packaging) in a contact-lens wearing population in the US, ages 18-65. Derived CLUE scores using Item Response Theory (IRT) follow a normal distribution with a population average score of 60 (SD 20), where higher scores indicate a more favorable/positive response with a range of 0-120. The average CLUE vision score for each lens type was reported.
Time Frame: 1-Week Follow-up
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Test (Senofilcon A C3) | Control (Delefilcon A)
Number analyzed (Participants) | 36 | 34
Units on a scale | 49.80 (19.662) | 52.35 (19.212)
Statistical Analysis 1: Comparison: Test (Senofilcon A C3); It was calculated using a 2-sided one sample mean t-test with a family wise type I error rate of 5% (1.25% individually) with at least 99% statistical power, that 13 subjects were required to test for superiority for CLUE vision scores; Test type: Superiority — Superiority was declared if the lower bound of the 98.75% confidence interval was above 32; Linear Mixed Model; Kenward and Roger method was used for denominator degrees of freedom; Least-square Mean = 50.8, 98.75% CI 2-sided [43.1 to 58.5], Standard Error of Mean 2.922

3. Secondary Outcome: Binocular Distance logMAR Visual Acuity
Description: Binocular visual acuity was measured on a logMAR (Logarithm of Minimal Angle of Resolution) scale at distance (4m) under high luminance high contrast condition assessed using ETDRS (Early Treatment Diabetic Retinopathy Study) charts. Letter-by-letter results calculated the visual performance score for each chart read. LogMAR scores closer to zero, or below zero, indicate a better visual acuity. A logMAR visual performance score of 0.0 is equivalent to Snellen visual acuity of 20/20.
Time Frame: 1-Week Follow-up
Population: All subjects that completed all study visits without a major protocol deviation.
Measure: Mean (Standard Deviation); unit: LogMAR
Arm/Group | Test (Senofilcon A C3) | Control (Delefilcon A)
Number analyzed (Participants) | 33 | 32
LogMAR | -0.078 (0.0942) | -0.083 (0.1080)
Statistical Analysis 1: Comparison: Test (Senofilcon A C3) vs Control (Delefilcon A); It was calculated using a 2 independent sample means t-test with a 2-sided type I error rate of 5% with at least 95% statistical power, that 60 subjects were required to test for non-inferiority of the Test compared to the Control for distance (4m); Test type: Non-Inferiority — Non-inferiority was declared if the upper limit of the 95% confidence interval of the least-square mean difference was below 0.05 logMAR; Linear Mixed Model; Kenward and Roger method was used for denominator degrees of freedom; LSM Difference = 0.00, 95% CI 2-sided [-0.05 to 0.05], Standard Error of Mean 0.024 — LSM difference was calculated as Test minus Control

ADVERSE EVENTS:
Time Frame: Throughout the duration of the study; The study duration for each subject was approximately 17±3 days.
Groups:
- Test (Senofilcon A C3): Subjects that wore the Control lens during the study.
- Control (Delefilcon A): Subjects that wore the Test lens during the study.
Arm/Group | Test (Senofilcon A C3) | Control (Delefilcon A)
All-Cause Mortality (participants affected / at risk) | 0/37 | 0/37
Serious Adverse Events (participants affected / at risk) | 0/37 | 0/37
Other Adverse Events (participants affected / at risk) | 0/37 | 0/37

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-09-29): https://cdn.clinicaltrials.gov/large-docs/52/NCT05101252/Prot_SAP_000.pdf